CLINICAL TRIAL: NCT01439113
Title: A Randomized Trial of Single-Operator Ultrasound-Guided vs. Standard-of-Care IV Placement by Emergency Nurses
Brief Title: Single-operator Ultrasound-guided IV Placement by Emergency Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: usivedrn
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Intravenous Infusions
Keywords: Ultrasound, Difficult access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (No Intervention): In this arm, patients who have difficult IV access will undergo the standard of care. The options include a) repeated attempts by a primary nurse, b) new attempts by a second nurse, c) central line placement by a physician, d) intraosseous line placement by a physician, e) physician use of ultrasound for peripheral IV placement
- Ultrasound-guided IV (Experimental): In this arm, the emergency nurse will apply the ultrasound machine to locate and cannulate a patient's peripheral veins
  Interventions: Procedure: Ultrasound guided IV placement

INTERVENTIONS:
Procedure: Ultrasound guided IV placement — The nurse will use the emergency department's ultrasound machine to locate peripheral veins and then cannulate the vessel under ultrasound guidance.
  Arms: Ultrasound-guided IV

SUMMARY:
The placement of peripheral intravenous lines (IVs) is central to the treatment of patients in the emergency department (ED). The procedure is used for phlebotomy and administration of a variety of therapeutic medications and intravenous fluids. This procedure is standard of care, and IVs are routinely placed by experienced emergency nurses.

Occasionally, the nurse will have difficulty placing an IV line. The most common reason for this is an underlying medical condition, such as diabetes, severe peripheral vascular disease, obesity, or a history of intravenous drug use. When a nurse is unable to place an IV, the options are:

1. Ask another nurse to attempt the line placement
2. Ask a physician to establish access, which usually involves placement of a central venous catheter, a time-consuming procedure with higher risk of infection than a peripheral line.

The use of bedside ultrasound has become commonplace in the modern ED, and the Tufts Medical Center ED possesses its own machine, which is used for a variety of indications including diagnosis of pregnancy, gall bladder disease, abdominal free fluid or pericardial effusion. Another key use of bedside ultrasound is the location of blood vessels. In fact, it is now expected that when placing a central venous catheter the clinician use ultrasound guidance, as the ultrasound clearly demonstrates blood vessels. The procedure is completely pain-free and harmless, and costs nothing to perform.

Recently, there has been a growing body of evidence demonstrating that placement of peripheral IVs can be facilitated by the use of ultrasound. Just as it is useful for central venous catheters, ultrasound can also clearly show smaller peripheral veins. Multiple studies have demonstrated that physicians can place IVs with ultrasound guidance.

However, nurses are the de facto experts at placing peripheral IVs as it is a usual procedure for them to perform and they perform the procedure multiple times a day. In this study, we will provide a two-hour training program to a cohort of nurses. The training program will instruct them in the use of single-operator ultrasound-guided IV placement. After training, once the nurse encounters a patient with difficult IV access (either 2 failed attempts or history of difficult access), the patient will be consented and randomized to either the standard of care (whatever the nurse elects to do) or use of the bedside ultrasound.

In the meantime, the research assistant will measure time to IV placement starting from enrollment, the number of skin punctures that are necessary to place the IV, and then ask the patient questions about satisfaction with the IV placement and the pain they experienced.

Our hypothesis is that single-operator, ED nurse use of bedside ultrasound will facilitate IV placement in patients with difficult IV access, saving time and also improving patient satisfaction and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Any patient in whom IV access is indicated but either a) have a history of difficult IV access (either by self-report or by knowledge of the nurse or physician) or in whom two unsuccessful attempts (defined as skin punctures) have failed.

Exclusion Criteria:

* Patients will be excluded who are intoxicated, have acute psychiatric illness with exacerbation, who are prisoners, who cannot provide consent for themselves and who do not speak English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Need for intervention by a physician to obtain IV access | 1 year
  The number of times a physician needs to intervene to place an IV when the nurse confronts a patient with difficult IV access

SECONDARY OUTCOMES:
Time to IV placement | 1 year
  The time it takes to obtain IV access
Patient pain perception | 1 year
  The pain (on a standard 0-10 scale) that a patient perceives when an IV is placed
Number of skin punctures required to obtain IV access | 1 year
  The number of skin punctures required to obtain IV access

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts